CLINICAL TRIAL: NCT04621396
Title: Genetic and Environmental Influences on Development of Type 2 Diabetes in Childhood: The Next Generation Longitudinal Birth Cohort.
Brief Title: The Next Generation Longitudinal Birth Cohort Diabetes Study
Acronym: NextGen
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Brandy Wicklow, Assistant Professor, Pediatrics and Child Health, University of Manitoba
Other Study IDs: H2013:227
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes; Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pregnant women: A1C, lipoprotein profile, adiponectin, leptin, apo A and B, AST, and ALT, and HNF1a status.
  Birth: HNF1a status, apo A and B, glucose, insulin, c-peptide, and free fatty acid, leptin, and adiponectin, c-reactive protein (CRP), cytokines (interleukins and TNF alpha) will be tested on infant cord blood. Kidney ultrasound will be done to see the size of the kidney.
  1 to 18: creatine, albumin measurements, and urinalysis will be collected every year. Starting at age 2 and every 2 years afterward, urine will be frozen to test for biomarkers that may predict kidney damage or uncover causes for kidney damage in the future.
  7 to 18: A1C, OGTT, glucose levels, insulin levels, apolipoprotein A and B, c-reactive protein, lipoprotein profile, ALT, AST, leptin, and adiponectin. Between age 7 and 18: A1C, OGTT, glucose levels will be collected biennially. Blood samples will be frozen to test for biomarkers involved in developing T2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Next Generation Cohort: We will follow the children from mothers who either have T2D, GDM, or are controls.
  Interventions: Other: Observational screening study

INTERVENTIONS:
Other: Observational screening study

SUMMARY:
The overall aim of this project is to understand the independent roles of maternal factors, intrauterine exposures, genetic factors, and postnatal environment on the development of obesity and youth-onset type 2 diabetes (T2D) in childhood.

DETAILED DESCRIPTION:
Our primary objective for the study is to clinically and metabolically phenotype parents and their offspring to identify risk factors for obesity, T2D, and cardiometabolic risk in childhood and adolescence in a prospective birth cohort by reporting:

1. Maternal and/or paternal factors including anthropometrics, metabolic parameters, HNF1a genotype, lifestyle (diet and physical activity), and socioeconomic environment.
2. Infant factors including anthropometrics, early infant nutrition, and metabolism.

Secondary Objectives:

1. To evaluate if children born to mothers with T2D prior o pregnancy are at increased risk of obesity and T2D.
2. To determine the modifiable risk factors which contribute to the increased risk of obesity and T2D.
3. To evaluate the differential risk between mothers and fathers with T2D in terms of somatic and genetic contributions to risk compared to intrauterine environmental contributions to risk.
4. To plan a large-scale, randomized, controlled community-based breastfeeding intervention with intensive breastfeeding counseling and support for the prevention of T2D development in offspring of mothers or fathers with youth onset T2D.
5. To explore potential new research questions and feasibility studies for epigenetic studies using cord blood under the umbrella of the new research theme on T2D at the Children's Hospital Research Institute of Manitoba.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with type 2 diabetes, gestational diabetes, or no diabetes.
* From self-identified Indigenous heritage (e.g., Cree, Oji-Cree, Métis, Anishinaabe, etc.).
* Are delivering and residing in Manitoba.
* Mother/Father and children must be biological family members.

Exclusion Criteria:

* Mothers or children with type 1 diabetes.
* Residing outside of Manitoba.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children between the age of 0 and 18 or until a diagnosis of type 2 diabetes.
  Diagnosis of diabetes will be made according to the Canadian Diabetes Association criteria. There must be 2 abnormal blood glucose tests on different days OR 1 abnormal blood glucose test + symptoms of diabetes:
  Fasting plasma glucose of > 7.0 mmol/L or Random glucose > 11.1mmol/L or 2-hour glucose > 11.1 mmol/L after a standard oral glucose tolerance test (75g).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Obesity | 18 years
  Development of obesity defined by the International task force on obesity cut offs for age and gender.
Type 2 Diabetes | 18 years
  Development of type 2 diabetes defined by diagnostic criteria in the Canadian Diabetes association 2008 guidelines in childhood (≤ 7 years) or adolescence (12-16 years).

CONTACTS AND LOCATIONS:
Overall Officials: Brandy A Wicklow, MD, MSc, Principal Investigator — University of Manitoba, Children's Hospital Research Institute of Manitoba
Locations (1):
- Children's Hospital Research Institute of Manitoba/University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendelson M, Cloutier J, Spence L, Sellers E, Taback S, Dean H. Obesity and type 2 diabetes mellitus in a birth cohort of First Nation children born to mothers with pediatric-onset type 2 diabetes. Pediatr Diabetes. 2011 May;12(3 Pt 2):219-28. doi: 10.1111/j.1399-5448.2010.00694.x. Epub 2011 Mar 23. PMID 21429061
- See also: Website that has all the current projects that deal with diabetes. — https://www.dreamdiabetesresearch.com/